CLINICAL TRIAL: NCT03756870
Title: REvascularization Versus Optimal Medical Therapy on Left Ventricular ISchemia Reduction: Exploring the Associations Between Ischemia, Functional Outcome and Collaterals in the Treatment of Chronic Total Occlusion Patients
Brief Title: Revascularization Versus Optimal Medical Therapy of Chronic Total Coronary Occlusions on Left Ventricular Ischemia Reduction
Acronym: REVISE-CTO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, J.P.S Henriques, Principal Investigator, Head of Catheterization Laboratory, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REVISE-CTO
Record Dates: First submitted 2018-11-26; First posted 2018-11-28 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: Chronic Total Occlusion of Coronary Artery
Keywords: Chronic total coronary occlusion; Percutaneous coronary intervention; Optimal medical therapy; Myocardial ischemia
MeSH Terms: conditions — Myocardial Ischemia | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Intervention Model Description: 1:1 parallel design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CTO PCI (Experimental): Patients will receive optimal medical therapy, with percutaneous coronary intervention of the chronic total occlusion.
  Interventions: Procedure: Percutaneous coronary intervention (PCI)
- OMT (No Intervention): Patients will receive optimal medical therapy, without percutaneous coronary intervention of the chronic total occlusion.

INTERVENTIONS:
Procedure: Percutaneous coronary intervention (PCI) — A percutaneous coronary intervention of the chronic total occlusion with a drug-eluting stent.
  Arms: CTO PCI

SUMMARY:
Rationale: Randomized trials could not yet establish favourable outcomes of CTO PCI on hard endpoints such as ejection fraction or mortality, when compared to optimal medical therapy. However, patients after CTO PCI appeared to be more frequently free of angina complaints, but the aetiology behind this is not fully understood. The investigators hypothesize that PCI of the CTO in patients preselected with an ischemic threshold (>12.5%) on cardiac imaging leads to a reduction of the ischemic burden and therefore an increased benefit on functional outcomes.

Objective: Primary objective is to determine whether PCI of the CTO will yield a higher reduction of ischemia assessed by exercise myocardial perfusion SPECT-CT from baseline to 6-month follow-up compared to a control group. Secondary objectives are 1) to evaluate the effect of PCI of the CTO on improvement in functional status, infarct size and left ventricular function from baseline to follow-up compared to the control group; 2) to study the association between ischemia reduction and functional outcome and left ventricular function; 3) to assess the influence of the collateral flow index on the ischemic burden (reduction), functional status, infarct size and left ventricular (contractile) function (hibernation).

Study design: open multicentre randomized trial

Study population: 82 patients eligible for CTO PCI

Intervention: CTO PCI

Primary endpoint: ischemic burden assessed with exercise myocardial perfusion SPECT-CT from baseline to 6 months follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. A chronic total occlusion is present and target lesion. A CTO is required to meet the following characteristics:

   * A 100% luminal narrowing of the coronary artery without antegrade flow, i.e. Thrombolysis in Myocardial Infarction flow grade 0 or 1;
   * Older than 3 months, established with previous PCI or with angiographic characteristics;
   * Amenable to percutaneous revascularization.
2. Patient has a clinical indication to perform CTO PCI.
3. A SPECT is performed at baseline to assess ischemia and a cardiac magnetic resonance imaging (CMR) scan to assess viability, as part of routine patient care. Patients are deemed eligible for the randomized trial when they meet the ischemic threshold in the CTO territory.

   The ischemic threshold is defined as:
   * >12.5% of ischemia;
   * With <50% transmural extent of infarction.
4. Subject agrees to undergo follow-up SPECT-CT at 6 months after initial inclusion
5. Subject is able to verbally confirm understanding and he/she provides written informed consent prior to any Clinical Investigation related procedure, as approved by the appropriate Ethics Committee.

Exclusion Criteria:

* Subject is younger than 18 years of age;
* Persistent or permanent atrial fibrillation;
* Presence of a non-MRI compatible cardiac device, i.e. pacemaker or implantable cardioverter defibrillator;
* Body weight > 250 kg;
* Unable to exert, i.e. due to physical disability;
* Any contraindication for SPECT or CMR, i.e. cerebrovascular clips, claustrophobia;
* Known renal insufficiency (estimated Glomerular Filtration Rate [eGFR] <60 mL/min/1.73m2 or serum creatinine level of >2.5 mg/dL or subject on dialysis);
* Hypersensitivity or allergy to contrast with inability to properly pre-hydrate;
* Presence of a comorbid condition with a life expectancy of less than one year;
* Participation in another trial;
* Subject is belonging to a vulnerable population (per investigator's judgment, e.g., subordinate hospital staff) or is unable to read or write.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Estimated)
Dates: Start 2019-07-01 (Actual); Primary Completion 2024-01-01 (Estimated); Study Completion 2030-01-01 (Estimated)

PRIMARY OUTCOMES:
Ischemia | 6 months follow-up
  Ischemic burden assessed with exercise myocardial perfusion SPECT-CT from baseline to 6 months follow-up.

SECONDARY OUTCOMES:
Change in angina status assessed with the Seattle Angina Questionnaire. | 6 months, 1 year, 2 years, 3 years, 4 years, 5 years, 6 years, 7 years, 8 years, 9 years, 10 years
  5 Seattle Angina Questionnaire subscales (0-100), higher scores indicating better angina status.
Quality of life assessed with the Minnesota Living with Heart Failure Questionnaire (MLHFQ) | 6 months, 1 year, 2 years, 3 years, 4 years, 5 years, 6 years, 7 years, 8 years, 9 years, 10 years
  MLHFQ scale (0-105), lower scores indicating better quality of life.
The left ventricular ejection fraction assessed with cardiac magnetic resonance imaging | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Amsterdam UMC, location AMC, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided